CLINICAL TRIAL: NCT05110560
Title: Effects of the "Stay at Home-Take a Step" Programme Developed for Sedentary Elderly in the COVID-19 Pandemic: Mobile Interventional Study
Brief Title: Effects of the Programme Developed for Sedentary Elderly in the COVID-19 Pandemic: Mobile Interventional Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Namik Kemal University (Other)
Responsible Party: Principal Investigator, Nurhan Ozpancar, Assistant Professor, Namik Kemal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Namik Kemal University
Record Dates: First submitted 2021-10-06; First posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Aged
Keywords: COVID 19; Elderly; Step Count; Walking
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: "Stay at Home Take a Step Program (SHTSP)" will be performed with the intervention group.
  For the control group, only the number of steps will be followed.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): step counts will be followed
- intervention group (Experimental): The Stay at Home Take a Step Program consisting of video or audio calls four times, sending Short Message Service messages containing reminders to encourage walking, and daily step count and weight tracking will be implemented.
  Interventions: Behavioral: "Stay at Home Take a Step Program (SHTSP)"

INTERVENTIONS:
Behavioral: "Stay at Home Take a Step Program (SHTSP)" — The Stay at Home Take a Step Program consisting of video or audio calls four times, sending Short Message Service messages containing reminders to encourage walking, and daily step count and weight tracking will be implemented.
  Arms: intervention group

SUMMARY:
The purpose of all these applications is the same: people keep distance and isolate themselves from those in risk groups and patients. In Turkey, it was announced by the Ministry of Health (2020) that the first official COVID-19 case was seen on March 11, 2020. Immediately afterwards, many pioneering measures were taken, such as travel restrictions, mandatory quarantine practices for those with a foreign history, interruption of primary, secondary and higher education, closure of common areas curfews. In order to minimize contact and ensure social isolation, home quarantine practice was encouraged with the 'Stay at Home Turkey' campaign. Within the scope of the measures taken, a curfew was imposed for citizens over 65 years of age who are considered to be risky in terms of high death rate and who have chronic diseases, as of 21 March - 9 June 2020, and the elderly population became the first group to leave social environments in our country. However, quarantine and social isolation for the elderly population due to increased sedentary lifestyle and loneliness pose a serious public health problem. The COVID-19 epidemic has affected health and quality of life in many ways, and one of the most affected areas has been healthy lifestyle behaviors.

Especially sedentary and sedentary life is of vital importance for the elderly. When the literature in this field is examined, it is shown that physical activity reduces the risk of premature death, supports positive mental health and supports healthy aging More importantly, physical activity sessions don't have to be long to improve health; 10-minute bouts of moderate to vigorous physical activity are beneficial for the prevention and control of diseases, and even light activity such as moderate-paced walking is beneficial. In addition, emphasized that walking is a low-cost activity that, if done at recommended levels, can reduce the incidence of chronic diseases and associated health care costs. No expensive equipment or gym membership required to walk; most people can do this by incorporating it into their daily life. In this study, which is planned from here, it is aimed to examine the effect of the stay at home program, which is carried out with the mobile initiative to gain exercise behavior in elderly individuals over the age of 65 who are under mandatory quarantine at their homes during the COVID 19 pandemic process, on the number of steps, quality of life and stress level.

DETAILED DESCRIPTION:
Type of Research The study was designed as a randomised controlled study with the control group Research Sample

The population of the study consists of individuals over the age of 65 in Turkey during the COVID 19 pandemic. For this purpose, information messages were sent to Tekirdag Namik Kemal University undergraduate students who continue their distance education between 15 May-1 June. The students were asked to invite individuals aged 65 and over who are in their immediate environment (relatives, neighbors, etc.) who meet the inclusion criteria to participate in the study. All volunteer participants in the determined date section were called by phone and their compliance with the inclusion and exclusion criteria was evaluated. All participants meeting the inclusion criteria were included in the study population (n= 94). If the minimum sample size cannot be reached, it is planned to extend the participation period in the study. The sample size was calculated using the G Power program to calculate the minimum number of samples to be used in the study. In determining the sample size, considering the previously published articles in which similar interventions were applied, Type 1 error amount was 0.05, test power was 0.95, and effect size: 0.83; The minimum number of samples required was determined as 64 (32 experimental + 32 control group) for the experimental and control groups. All participants meeting the inclusion criteria were randomly divided into experimental and control groups by a statistician outside the study using the Random Online Allocation Software program (www.Graphpad.com). A double-blind technique was used in the assignment of the groups.

Research Process After obtaining the ethics committee and institutional permissions for the research, "Socio-demographic information form", "EuroQOL General Quality of Life Scale" and "Perceived Stress Scale" online questionnaires were applied to all elderly people who met the inclusion criteria as a pre-test. Elderly people who have vision problems and could not answer the online questionnaire were asked to read and answer questions by telephone interview. In addition, a pedometer device was sent to all the elderly in the experimental and control groups. It will be explained in detail how to use it, and they will be asked to record the number of steps and weights on the "Following Chart" for 2 months. Unlike the control group, the intervention group will be applied to the "Stay at Home Step by Step Program" (EKAAP), which will last for 4 weeks.

As a post-test, "Socio-demographic information form", "EuroQOL General Quality of Life Scale" and "Perceived Stress Scale" will be applied to both the experimental and control groups. One month after the intervention is completed, it will be possible to monitor the change in step counts, weight values, EuroQOL General Quality of Life Scale and Perceived Stress Scale scores of the elderly.

Data Collection Tools

1. Socio-Demographic Information Form The Descriptive Questionnaire was created by the researchers by examining the relevant literature. This form includes questions about socio-demographic characteristics (age, marital status, gender, education level, number of children, people with whom they live, place of residence, household size, employment status).
2. EuroQOL General Quality of Life Scale It is a scale developed to assess health-related quality of life. It consists of two parts: Chapter 1 defines the health profile in five dimensions (mobility, self-care, social life, pain and psychological state). Each dimension contains three statements according to difficulty (1 a little problem; 2 medium; 3 a lot of problems), Section 2 includes the visual analog scale, in which respondents rate their current health status on a scale of 0 to 100. Easy to apply and quickly identified.Turkish validity and reliability were done by Kahyaoglu Süt and Ünsar.
3. Perceived Stress Scale The scale was developed by Cohen et al. Its validity and reliability study was conducted by Erci, and it was determined that it was adapted to Turkish society and appropriate.The scale consists of 10 items, and each item receives 1, 2, 3, 4, 5 points, respectively.The scale is evaluated over the total score and the scores are calculated between 10-50. A score of 30 and above indicates that the individual has stress. As the score increases, the stress level also increases. In the validity and reliability study of the scale, it was determined that the test-retest correlation was 0.88.

Statistical procedure

Percentage, mean, standard deviation will be used in the evaluation of the data. Chi-square, Fisher's exact test, independent paired T-test and Mann-Whitney U test will be used for comparison between groups and within groups. p <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Those who volunteered to participate in the study
* No mental disability,
* Can read and write Turkish
* Using a smartphone
* No muscle-joint problems that interfere with physical activity
* No neuropsychiatric disorder
* No cognitive problem that prevents communication
* Not diagnosed as COVID 19 positive
* Able to carry out activities of daily living independently
* All individuals aged 65 and over will be included. Sedentary elderly people who take an average of 2000 or less steps per day

Exclusion Criteria:

* Having insulin-dependent Type 2 diabetes
* Having hypertension and not being able to control it with medication
* Being diagnosed with Heart Failure
* Being diagnosed with chronic obstructive pulmonary disease
* Being diagnosed with asthma
* Being diagnosed with cancer

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Daily steps | from the start of the study to the first month
  Daily walking amount will be assessed by number of steps/day. The number of steps of the participants will be measured and recorded with the pedometer device.
  The sedentary elderly who took an average of 2000 or less steps per day were included in the study.
EuroQoL Quality of Life Scale | after attempt completion and one month later
  Quality of Life will be assessed by EuroQoL Quality of Life Scale total point. Scale consists of two parts: Part 1 defines the health profile in five dimensions. Each dimension contains three statements according to difficulty (1 some problem; 2 moderate; 3 a lot of problems), part 2 includes a visual analog scale where respondents rate their current state of health on a scale of 0 to 100.
Stress level | after attempt completion and one month later
  Stress level will be assessed by Perceived Stress Scale total point. Perceived Stress Scale is evaluated over the total score and the scores are calculated between 10-50. A score of 30 and above indicates that the individual has stress. As the score increases, the stress level also increases.

CONTACTS AND LOCATIONS:
Overall Officials: NURHAN ÖZPANCAR, Principal Investigator — Namik Kemal University; AYLİN YALÇIN IRMAK, Principal Investigator — Namik Kemal University
Locations (1):
- Namik Kemal University, Tekirdağ, Süleymanpasa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sipila S, Tirkkonen A, Hanninen T, Laukkanen P, Alen M, Fielding RA, Kivipelto M, Kokko K, Kulmala J, Rantanen T, Sihvonen SE, Sillanpaa E, Stigsdotter-Neely A, Tormakangas T. Promoting safe walking among older people: the effects of a physical and cognitive training intervention vs. physical training alone on mobility and falls among older community-dwelling men and women (the PASSWORD study): design and methods of a randomized controlled trial. BMC Geriatr. 2018 Sep 15;18(1):215. doi: 10.1186/s12877-018-0906-0. PMID 30219032
- [Result] Branco JC, Jansen K, Sobrinho JT, Carrapatoso S, Spessato B, Carvalho J, Mota J, da Silva RA. Physical benefits and reduction of depressive symptoms among the elderly: results from the Portuguese "National Walking Program". Cien Saude Colet. 2015 Mar;20(3):789-95. doi: 10.1590/1413-81232015203.09882014. PMID 25760119
- [Result] Rye Hanton C, Kwon YJ, Aung T, Whittington J, High RR, Goulding EH, Schenk AK, Bonasera SJ. Mobile Phone-Based Measures of Activity, Step Count, and Gait Speed: Results From a Study of Older Ambulatory Adults in a Naturalistic Setting. JMIR Mhealth Uhealth. 2017 Oct 3;5(10):e104. doi: 10.2196/mhealth.5090. PMID 28974482